CLINICAL TRIAL: NCT05103501
Title: Salvage Immunotherapy Combined With Chemotherapy in Esophageal Squamous Cell Carcinoma Patients Nonresponding to Initial Neoadjuvant Chemoradiotherapy (SINCERE Study)
Brief Title: Salvage Immunotherapy and Chemotherapy in Esophageal Squamous Cell Carcinoma Patients Nonresponding to Initial Neoadjuvant Chemoradiotherapy
Acronym: SINCERE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Jun Liu, associate proffessor, Shanghai Chest Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JLiu
Record Dates: First submitted 2021-10-11; First posted 2021-11-02 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Esophageal Squamous Cell Carcinomas
MeSH Terms: interventions — CF regimen; Cisplatin; Fluorouracil

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental arm (Experimental): PF regimen (cis-platinum of 75mg/m2/d, d1; 5-fluorouracil of 600mg/m2d1-4) combined with PD-1 inhibitors（pembrolizumab，200mg d1） every 3 weeks for 4 cycles followed by PD-1 inhibitors（pembrolizumab，200mg d1）every 3 weeks up to 2 years in a standard manner.
  Interventions: Drug: PF regimen (cis-platinum ; 5-fluorouracil ) combined with PD-1 inhibitors（pembrolizumab）

INTERVENTIONS:
Drug: PF regimen (cis-platinum ; 5-fluorouracil ) combined with PD-1 inhibitors（pembrolizumab） — immunotherapy:PD-1 inhibitor chemotherapy:5-Fu and DDP

SUMMARY:
This is an investigator-initiated, single-arm, exploratory clinical study.The study population consisted of esophageal squamous cell carcinoma patients nonresponding to initial neoadjuvant chemoradiotherapy. The purpose of this study was to evaluate the efficacy and safety of immunotherapy combined with chemotherapy in the adjuvant treatment of esophageal squamous cell carcinoma after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with Stage II/III carcinoma of the esophagus squamous cell carcinoma.
2. Completed pre-operative chemoradiotherapy followed by surgery
3. Diagnosed with residual pathologic disease after being surgically rendered free of
4. Disease with negative margins following complete resection
5. Nonresponding to initial neoadjuvant Chemoradiotherapy(TRG3 and TRG4)

Exclusion Criteria:

1. Known or suspected history of active autoimmune diseases, autoimmune diseases (such as interstitial pneumonia, colitis, hepatitis, pituitaritis, vasculitis, nephritis, hyperthyroidism, hypothyroidism, including but not limited to these diseases or syndromes)
2. Have a history of immunodeficiency, including HIV positive, or other acquired, congenital immunodeficiency disease, or history of organ transplantation and bone marrow transplantation；
3. Interstitial lung disease, drug-induced pneumonia, radiation pneumonitis requiring steroid therapy or active pneumonia with clinical symptoms or severe pulmonary dysfunction；
4. There are clinical symptoms or diseases of the heart that are not well controlled, such as: (1) heart failure of NYHA class 2 or higher (2) unstable angina (3) myocardial infarction within 24 weeks (4) clinical need for treatment or Interventional supraventricular or ventricular arrhythmia；
5. Have a tendency to hereditary bleeding or coagulopathy. Clinically significant bleeding symptoms or clear bleeding tendency within 3 months prior to enrollment, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, baseline fecal occult blood++ and above；
6. Has not fully recovered from toxicity and/or complications from any intervention prior to initiation of treatment (i.e., ≤ grade 1 or level required at baseline, excluding fatigue or hair loss);
7. Allergic reactions to test drugs for this application；
8. Pregnant or lactating women； Those whom the investigator considered unsuitable for inclusion。

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Disease-free Survival (DFS) | up to approximately 46 months
  Disease-free survival is defined as the time between date of surgery and first date of recurrence or death, whichever occurs first.Recurrence is defined as the appearance of one or more new lesions, which can be local, regional, or distant in location from the primary resected site ( assessed by imaging or pathology). All deaths without prior recurrence are considered as DFS events.

SECONDARY OUTCOMES:
Overall survival (OS) | up to approximately 46 months
  Overall survival is defined as the time from date of surgery to date of death from any cause. For subjects that are alive, their survival time was censored at the date of last contact date (or "last known alive date").
Overall Survival Rate | From date of surgery to 1, 2 and 3 years later
  Overall survival rate is defined as the percentage of participants who are alive at 1, 2 and 3 years following surgery

IPD SHARING:
Plan to Share IPD: No